CLINICAL TRIAL: NCT03832426
Title: An Open Label, Parallel Design Study to Assess the Pharmacokinetics of Narlaprevir 200 mg as a Single Oral Dose and in Combination With Ritonavir 100 mg in Patients With Hepatic Impairment and Healthy Matched Volunteers
Brief Title: A Pharmacokinetic Study of Narlaprevir as a Single Dose or With Ritonavir Combination in Patients With Hepatic Impairment and Healthy Matched Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Ascent (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJ05013007
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — narlaprevir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Narlaprevir single - Healthy (Experimental): 2 tablets of 100 mg Narlaprevir once a day
  Interventions: Drug: Narlaprevir
- Narlaprevir single - Hepatic Impairment (Experimental): 2 tablets of 100 mg Narlaprevir once a day
  Interventions: Drug: Narlaprevir
- Narlaprevir+Ritonavir - Healthy (Experimental): Narlaprevir 100 mg (1 tablet of 100 mg) and Ritonavir 100 mg (1 tablet of 100 mg) once a day
  Interventions: Drug: Narlaprevir; Drug: Ritonavir
- Narlaprevir+Ritonavir - Hepatic Impairment (Experimental): Narlaprevir 100 mg (1 tablet of 100 mg) and Ritonavir 100 mg (1 tablet of 100 mg) once a day
  Interventions: Drug: Narlaprevir; Drug: Ritonavir

INTERVENTIONS:
Drug: Narlaprevir — 100 mg film-coated tablets
Drug: Ritonavir — 100 mg film-coated tablets
  Arms: Narlaprevir+Ritonavir - Healthy; Narlaprevir+Ritonavir - Hepatic Impairment

SUMMARY:
This study was conducted to evaluate narlaprevir (NVR) pharmacokinetics (PK) after a single dose with or without ritonavir (RTV) in cirrhotic Child-Pugh class A patients without active HCV infection versus healthy subjects as well as to assess safety and tolerability of such treatment combination.

DETAILED DESCRIPTION:
The objective of this study was to evaluate PK after a single oral dose of NVR alone and in combination with RTV in patients with compensated liver cirrhosis and in matched healthy controls.

The study consisted of 2 parts. In Part I of the study, 8 patients with compensated cirrhosis (Child-Pugh Class A) and 8 matched healthy adult subjects received single doses of NVR at 200 mg with 240 ml of water after a standard breakfast. The 200-mg NVR dose was chosen since this is the intended therapeutic dose. Blood and urine samples were obtained to determine narlaprevir concentration in plasma and urine.

As an additional safety precaution, patients with Child-Pugh Class A hepatic impairment were studied successively in Part I and Part II on the basis of the results of an interim safety analysis data and PK data.

Based on the results of the interim analysis after the Part I of the study, it was decided to reduce the dose of narlaprevir from baseline 200 mg to 100 mg in Part II of the study.

In part 2 of the study, 8 patients with compensated cirrhosis (Child-Pugh Class A) and 8 healthy subjects received NVR at 100 mg in combination with RTV at 100 mg with 240 ml of water after a standard breakfast. Blood and urine samples were obtained to determine narlaprevir concentration, its metabolite and ritonavir in plasma and urine.

The total duration of the study for each subject was a maximum of 35 days.

ELIGIBILITY:
Inclusion Criteria:

1. Common for patients and volunteers:

   * The study patient/volunteer could understand and fulfill the requirements of the Protocol (according to the Investigator)
   * The patient/volunteer signed and dated a written informed consent form and any other required permits for use of personal information prior to any study procedures.
   * The study subject was a healthy adult man or woman (for inclusion in the group of healthy volunteers) or had Child-Pugh Class A hepatic impairment (for inclusion in the group with hepatic impairment).
   * At screening, females capable of child-bearing had the result of a pregnancy test (β-hCG in blood plasma) corresponding to the absence of pregnancy and agreed to use adequate contraception during the study, starting at least 2 weeks prior to drug administration and the onset of menarche, but at least 2 weeks after drug administration; or passed the surgical sterilization at least 3 months prior to the study.
   * Menopausal females could participate in the study if they had no menstruation for at least 1 year and had the appropriate age. Menopausal status was confirmed in the screening by the appropriate level of FSH.
   * Males who were not surgically sterilized had to agree to use reliable methods of contraception after signing a consent form for the study for 90 days after administration of the study drug administration.
   * The study patient/volunteer was ready to refrain from caffeine and alcohol for the period from 72 hours prior to obtaining a dose of the study drug (Day 1) and until the final visit.
   * The study patient/volunteer was ready to refrain from excessive physical activity for the period from 72 hours prior to obtaining a dose of the study drug (Day 1) and until the final visit.
   * The body weight of study patient/volunteer at screening and on Day 1 was not less than 45 kg, and body mass index (BMI) - from 18.0 to 35.0 kg/m2, inclusive. BMI was calculated by dividing body weight of patient/volunteer in kilograms by the square of their height in meters.
   * The study patient/volunteer had no clinically significant abnormalities on the electrocardiogram (ECG) (QTc interval ≤450 msec in males and ≤470 msec in females) performed at the screening visit and before administration of the study drug on Day 1.
   * The study patient/volunteer agreed not to take the use of grapefruit or products containing them for the period of at least 2 weeks prior to the study drug administration until the end of the study. It was forbidden to drink any fruit juice for the period from 24 hours before narlaprevir administration until the end of the period of collecting the samples for pharmacokinetic analysis.
   * The study patient/volunteer agreed to refrain from the use of St. John's wort and products containing them and/or any other herbal medicines, organic and homeopathic medicines, dietary or nutritional supplements of any kind (except multivitamin drugs prescribed 1 per day) for at least 2 weeks prior to dosing and throughout the study.
   * The study patient/volunteer understood the study procedures and confirmed consent to participate therein by signing a consent form.
   * The study patient/volunteer was ready to provide a blood sample for pharmacogenetic analysis (optional).
2. Specific inclusion criteria for patients with hepatic impairment:

   * Evaluation of patient's liver function corresponds to 5-6 (mild hepatic insufficiency) on Child-Pugh scale at the screening visit.
   * On the basis of history, physical examination, vital signs and laboratory safety tests carried out at the screening visit and/or before the study drug administration, the patient did not have clinically significant diseases in addition to the existing liver failure. Patients with the test results outside the normal range that the Investigator considered clinically insignificant could have been included in the study on the discretion of the Investigator if it was not otherwise mentioned in the non-inclusion criteria.
   * The patient was diagnosed with chronic (> 6 months ago), stable (in previous 2 months did not have periods of acute illness due to deterioration of liver function) liver failure.
3. Specific inclusion criteria for the corresponding healthy volunteers:

   * A volunteer weighing ±10% from the parameter of the body weight corresponding to his/her patient with hepatic impairment included in the study.
   * A volunteer was recognized as healthy on the basis of history, physical examination, vital signs and laboratory safety tests carried out at the screening visit and/or before the study drug administration (Day 1).
   * A volunteer of the same race as the corresponding to his/her included patient with hepatic impairment.
   * A volunteer of the same gender as the corresponding to his/her included patient with hepatic impairment.
   * The age of a volunteer was within ±10 years from the age of the corresponding to his/her included patient with hepatic impairment.

Exclusion Criteria:

1. General criteria for exclusion of patients/volunteers:

   * A minor, mentally or legally incompetent patient/volunteer with a significant emotional disturbance at the screening visit, or those patients/volunteers who were assumed to have the development of such disorders during the study, or those who had a history of clinically significant mental disorders.
   * A patient/volunteer received any other study drug within 90 days prior to receiving the study drug dose.
   * A patient/volunteer received narlaprevir in a previous clinical study, or as a means for treating the disease.
   * A patient/volunteer had hypersensitivity to any component of narlaprevir or related substances.
   * A patient/volunteer had a positive urine test for prohibited drugs at the screening visit and on Day -1.
   * History of drug dependence of a patient/volunteer (defined as the use of any drug for entertainment) or alcoholism, or excessive drinking during the last year. Excessive drinking defined as consumption per week on average over 14 (for females) and 21 (for males) of alcoholic units (1 unit of alcohol = 8-10 g of alcohol and equivalent to about 200 ml of wine or 250 ml of beer, or standard measures for strong alcoholic beverages).
   * A patient/volunteer consumed excessive amounts of coffee, cola, tea or other caffeine-containing drinks per day. Excessive drinking was considered more than 6 servings (1 serving or about 120 mg of caffeine) per day.
   * A patient/volunteer received drugs, food supplements or food products prohibited in the study, with the exception of non-prescription drugs pre-approved for use by the Sponsor. When deciding on inclusion in the study, particular attention was paid to the use of such drugs as azole antifungals (ketoconazole, itraconazole), antibiotics, macrolides (erythromycin, clarithromycin), cimetidine, HIV protease inhibitors, nefazodone, rifampin, phenytoin, dexamethasone, troglitazone, barbiturates or any inducers or inhibitors of enzymes P-450 CYP3A or CYP2C9 and substrates or inhibitors of transport protein P-gp. In addition, drugs known under strong evidence for their ability to prolong the QT interval and cause polymorphic ventricular tachycardia should also have been considered as drugs of concern at inclusion.
   * Pregnant and lactating females as well as females who planned to become pregnant or to deliver eggs for fertilization before, during, or within 1 month after taking part in the study. The males who planned to deliver sperm for fertilization during the study or within 12 weeks after it.
   * A patient/volunteer had cancer in history other than basal cell carcinoma being in remission for at least 5 years before Day 1.
   * At screening, a patient/volunteer had positive results of tests for surface antigen of hepatitis B virus (HBsAG), for antibodies to hepatitis C virus (HCV), for antigen/antibody to human immunodeficiency virus (HIV). Patients/volunteers with hepatitis B or C in history were not included in the study. The study could include patients/volunteers with a history of hepatitis A from which they recovered without any treatment, if there was no documentary evidence on complete resolution of the disease for at least 6 months prior to Day 1.
   * A patient/volunteer underwent surgery, donated or lost 450 or more ml of blood (including plasmapheresis, or underwent transfusion of blood products within 90 days prior to Day 1.
   * A patient/volunteer had a history of gastroesophageal reflux disease (GERD), eosinophilic esophagitis, duodenal ulcer, gastric ulcer, dyspepsia, Barrett's esophagus or Zollinger-Ellison syndrome, or had a history of or had at the time of the study (during 6 months before screening) gastrointestinal diseases that could conceivably affect the absorption of drugs.
   * A history of strokes, seizures or severe chronic neurological disorders.
   * A patient/volunteer had a history of or had at the time of the study clinically significant endocrine, gastrointestinal, cardiovascular, hematologic, immune, renal, respiratory or urinary disorders or diseases which the Investigator believed to affect the correct evaluation of the study or pose additional risks to a patient/volunteer's participation in the study.
   * A patient/volunteer had creatinine clearance <60 ml/min under Cockcroft-Gault calculation at screening.
   * A patient/volunteer had multiple and/or severe allergy history or had a history of anaphylactic reactions or intolerance of certain prescription or nonprescription drugs or food.
   * At the time of selection, a patient/volunteer regularly consumed any illicit drugs (including those for entertainment) or had a history of drug or alcohol addiction for about 2 years.
   * The Investigator had any concerns about safety of a patient/volunteer participation in the study, or any other reason why the Investigator believed that the patient was not suitable for participation in the study.
   * A patient/volunteer was not able to refrain from the use or intended use of any prescription or non-prescription drugs or herbal preparations (for example, St. John's wort [hypericum perforatum], green tea, ginkgo, coenzyme Q, ginseng, Echinacea, etc.) or dietary supplements (e.g., garlic supplements) starting about 2 weeks (or 5 half-lives) before the study drug dosing throughout the study and before and before the visit after the study. Patients with hepatic impairment administered with medication for treatment of this disease could participate in the study, if these drugs were administered at stable state for at least 4 weeks.
2. Specific non-inclusion criteria for healthy volunteers:

   * A volunteer had a history of any chronic and/or acute liver disease, including an increase in transaminase serum levels, hepatitis, biliary tract disease, or a history of significant surgery on the gastrointestinal tract. The study could include volunteers who had a history of transient increase in transaminase levels fully resolved not later than 6 months before entering the study.
   * Any laboratory parameter exceeding ULN at screening visit established by the testing laboratory (if the deviation was considered clinically insignificant by the Investigator, the deviation could be ±10% from the normal range).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2014-10-24 (Actual); Study Completion 2014-10-24 (Actual)

PRIMARY OUTCOMES:
AUC (0-last) of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the area under the concentration-time curve from the time of dosing (time 0) before the observation time of the last detectable concentration
AUC (0-24) of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 hours after dosing
  area under the concentration-time curve from time 0 to 24 hours
AUC (0-48) of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48 hours after dosing
  the area under the concentration-time curve from time 0 to 48 hours
AUC (0-inf) of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the area under the concentration-time curve from time 0 to the time extrapolated to infinity
Cmax of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the maximum observed plasma concentration
Tmax of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the time to reach Cmax
t1/2 of Narlaprevir | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  terminal half-life

SECONDARY OUTCOMES:
Cu(t1-t2) of Narlaprevir | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  concentration of the drug excreted in the urine from time 1 to time 2
Vu(t1-t2) | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  urine volume, excreted from time 1 to time 2
Ae (0-t) | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  total amount of the drug excreted in the urine from time 0 to t
Ae (0-24) | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  total amount of the drug excreted in the urine from time 0 to 24 hours
Fe | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  drug fraction excreted in the urine
CLr | before dosing, 0-4, 4-8, 8-12, 12-16 and 16-24 hours after dosing
  renal clearance

OTHER OUTCOMES:
AUC (0-last) of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the area under the concentration-time curve from the time of dosing (time 0) before the observation time of the last detectable concentration
AUC (0-24) of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24 hours after dosing
  area under the concentration-time curve from time 0 to 24 hours
AUC (0-48) of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48 hours after dosing
  the area under the concentration-time curve from time 0 to 48 hours
AUC (0-inf) of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the area under the concentration-time curve from time 0 to the time extrapolated to infinity
Cmax of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the maximum observed plasma concentration
Tmax of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  the time to reach Cmax
t1/2 of Narlaprevir unbound fraction in plasma | before drug administration and in 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 36, 48, 72, 96 and 120 hours after dosing
  terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (3):
- Georgia (2):
  - LLC Chapidze Emergency Cardiology Center, Tbilisi
  - LLC Guli (Heart) - Cardiology clinic, Tbilisi
- - Institution of the Russian Academy of Sciences "RAS Hospital", Troitsk, Russia

REFERENCES:
- [Result] Isakov V, Koloda D, Tikhonova N, Kikalishvili T, Krasavina E, Lekishvili K, Malaya I, Ryska M, Samsonov M, Tolkacheva V. Pharmacokinetics of the New Hepatitis C Virus NS3 Protease Inhibitor Narlaprevir following Single-Dose Use with or without Ritonavir in Patients with Liver Cirrhosis. Antimicrob Agents Chemother. 2016 Nov 21;60(12):7098-7104. doi: 10.1128/AAC.01044-16. Print 2016 Dec. PMID 27645244